CLINICAL TRIAL: NCT04463290
Title: Association of Single Nucleotide Polymorphisms (SNPs) in Metalloproteinases (MMPs) Genes With the Risk of Primary Knee Osteoarthritis in Greek Population.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Christos Milaras, Orthopaedic Surgeon, Phd Candidate, Aristotle University Of Thessaloniki
Other Study IDs: 197/17.6.2020
Record Dates: First submitted 2020-07-05; First posted 2020-07-09 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Metalloproteinase SNPs -1575 G/A MMP-2, 836 A/G MMP-9 and -77 A/G MMP-13 and Risk for Developing Knee Osteoarthritis in Greek Population
Keywords: MMPs , SNPs, Knee osteoarthritis, -1575G/A MMP-2 , 836A/G MMP-9 , -77A/G MMP-13
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2ml blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Knee Osteoarthritis Patients Group: Patients suffering from primary knee osteoarthritis
  Interventions: Other: No intervention, Patients selection based on clinical symptoms and radiological imaging
- Control Group: Healthy people without suffering from primary knee osteoarthritis
  Interventions: Other: No intervention, Patients selection based on clinical symptoms and radiological imaging

INTERVENTIONS:
Other: No intervention, Patients selection based on clinical symptoms and radiological imaging — No intervention

SUMMARY:
Does the presence of gene polymorphisms -1575G / A in the MMP-2 gene, 836A / G in the MMP-9 gene and -77A / G in the MMP-13 gene, affect the risk of developing idiopathic knee osteoarthritis in the Greek population?

DETAILED DESCRIPTION:
This is a prospective case-control study in which the patients' genotype will be studied against the genotype of the controls. The study is prospective and not retrospective, as data will be collected from patients with primary knee osteoarthritis as well as the control group from the outset. The study intends to include 200 people. The first group consists of 100 individuals suffering from knee osteoarthritis, while the second group will include 100 healthy controls without osteoarthritis. From each one DNA will be isolated and analyzed from collected blood. The prospective study allows valid data to be collected on patient demographics and disease severity. Due to the large number of cases of the disease, it is estimated that the necessary specimens will be collected within a reasonable time from the beginning of this thesis. The choice of the patient-control study is necessary to limit the influence of confounding factors (age, gender, obesity, etc.). This type of study includes rigorous selection of patients and controls with specific entry and exclusion criteria, selection of controls based on matching patient characteristics, stratification, and subgroup analyzes. The final result will be a comparison of the incidence of specific gene polymorphisms between patients with knee osteoarthritis and the normal population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary knee osteoarthritis are selected based on clinical symptoms and radiological imaging with a score at least 2 on the Kellgren & Lawrence scale.
* Patients without symptomatology or radiographic image of knee osteoarthritis (score <2 on Kellgren & Lawrence scale) will be selected as controls.

Exclusion Criteria:

* systemic inflammatory disease
* rheumatic disease
* liver disease
* renal failure
* neoplasm or other chronic disease

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will take place at the 3rd Orthopedic Department of Aristotle University of Thessaloniki of the Papageorgiou General Hospital of Thessaloniki. The patients group will be patients with primary knee osteoarthritis coming for first examination for knee pain or for sceduled total knee arthroplasty surgery. The control group will be people coming for examination due to accident (trauma, fracture) or anything else not relevant with knee pain. Both groups must not have any of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-11-28 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The frequency of presence of gene polymorphisms -1575G / A MMP-2 gene, 836A / G MMP-9 gene and -77A / G MMP-13 gene, in Greek patients with knee osteoarthritis comparing with healthy people | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eleftherios Tsiridis, Professor, Study Director — Aristotle University of Thessaloniki, 3rd Orthopaedic Department, Medical School
Locations (1):
- 3rd Orthopedic Department , Pagageorgiou Hospital, Thessaloniki, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
The data that will be shared will be all the demographic data of the participants (gender, age, etc.) and the study results data. Personal participants data as name, address, telephone number will not be shared for any reason.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 12 months after publication
Access Criteria: Investigators from Greece, after personal contact.

REFERENCES:
- [Background] Shi J, Son MY, Yamada S, Szabova L, Kahan S, Chrysovergis K, Wolf L, Surmak A, Holmbeck K. Membrane-type MMPs enable extracellular matrix permissiveness and mesenchymal cell proliferation during embryogenesis. Dev Biol. 2008 Jan 1;313(1):196-209. doi: 10.1016/j.ydbio.2007.10.017. Epub 2007 Oct 23. PMID 18022611
- [Background] Hattori N, Mochizuki S, Kishi K, Nakajima T, Takaishi H, D'Armiento J, Okada Y. MMP-13 plays a role in keratinocyte migration, angiogenesis, and contraction in mouse skin wound healing. Am J Pathol. 2009 Aug;175(2):533-46. doi: 10.2353/ajpath.2009.081080. Epub 2009 Jul 9. PMID 19590036
- [Background] Salo T, Makela M, Kylmaniemi M, Autio-Harmainen H, Larjava H. Expression of matrix metalloproteinase-2 and -9 during early human wound healing. Lab Invest. 1994 Feb;70(2):176-82. PMID 8139259
- [Background] Duerr S, Stremme S, Soeder S, Bau B, Aigner T. MMP-2/gelatinase A is a gene product of human adult articular chondrocytes and is increased in osteoarthritic cartilage. Clin Exp Rheumatol. 2004 Sep-Oct;22(5):603-8. PMID 15485014
- [Background] Vu TH, Shipley JM, Bergers G, Berger JE, Helms JA, Hanahan D, Shapiro SD, Senior RM, Werb Z. MMP-9/gelatinase B is a key regulator of growth plate angiogenesis and apoptosis of hypertrophic chondrocytes. Cell. 1998 May 1;93(3):411-22. doi: 10.1016/s0092-8674(00)81169-1. PMID 9590175
- [Background] Soder S, Roach HI, Oehler S, Bau B, Haag J, Aigner T. MMP-9/gelatinase B is a gene product of human adult articular chondrocytes and increased in osteoarthritic cartilage. Clin Exp Rheumatol. 2006 May-Jun;24(3):302-4. PMID 16870098
- [Background] Dreier R, Grassel S, Fuchs S, Schaumburger J, Bruckner P. Pro-MMP-9 is a specific macrophage product and is activated by osteoarthritic chondrocytes via MMP-3 or a MT1-MMP/MMP-13 cascade. Exp Cell Res. 2004 Jul 15;297(2):303-12. doi: 10.1016/j.yexcr.2004.02.027. PMID 15212936
- [Background] Zeng GQ, Chen AB, Li W, Song JH, Gao CY. High MMP-1, MMP-2, and MMP-9 protein levels in osteoarthritis. Genet Mol Res. 2015 Nov 23;14(4):14811-22. doi: 10.4238/2015.November.18.46. PMID 26600542
- [Background] Shiomi T, Lemaitre V, D'Armiento J, Okada Y. Matrix metalloproteinases, a disintegrin and metalloproteinases, and a disintegrin and metalloproteinases with thrombospondin motifs in non-neoplastic diseases. Pathol Int. 2010 Jul;60(7):477-96. doi: 10.1111/j.1440-1827.2010.02547.x. PMID 20594269
- [Background] Li H, Wang D, Yuan Y, Min J. New insights on the MMP-13 regulatory network in the pathogenesis of early osteoarthritis. Arthritis Res Ther. 2017 Nov 10;19(1):248. doi: 10.1186/s13075-017-1454-2. PMID 29126436
- [Background] Harendza S, Lovett DH, Panzer U, Lukacs Z, Kuhnl P, Stahl RA. Linked common polymorphisms in the gelatinase a promoter are associated with diminished transcriptional response to estrogen and genetic fitness. J Biol Chem. 2003 Jun 6;278(23):20490-9. doi: 10.1074/jbc.M211536200. Epub 2003 Mar 25. PMID 12657623
- [Background] Beber AR, Polina ER, Biolo A, Santos BL, Gomes DC, La Porta VL, Olsen V, Clausell N, Rohde LE, Santos KG. Matrix Metalloproteinase-2 Polymorphisms in Chronic Heart Failure: Relationship with Susceptibility and Long-Term Survival. PLoS One. 2016 Aug 23;11(8):e0161666. doi: 10.1371/journal.pone.0161666. eCollection 2016. PMID 27551966
- [Background] Hua Y, Song L, Wu N, Xie G, Lu X, Fan X, Meng X, Gu D, Yang Y. Polymorphisms of MMP-2 gene are associated with systolic heart failure prognosis. Clin Chim Acta. 2009 Jun 27;404(2):119-23. doi: 10.1016/j.cca.2009.03.030. Epub 2009 Mar 28. PMID 19332048
- [Background] Morgan AR, Han DY, Thompson JM, Mitchell EA, Ferguson LR. Analysis of MMP2 promoter polymorphisms in childhood obesity. BMC Res Notes. 2011 Jul 21;4:253. doi: 10.1186/1756-0500-4-253. PMID 21777433
- [Background] Mossbock G, Weger M, Faschinger C, Zimmermann C, Schmut O, Renner W, El-Shabrawi Y. Role of functional single nucleotide polymorphisms of MMP1, MMP2, and MMP9 in open angle glaucomas. Mol Vis. 2010 Aug 28;16:1764-70. PMID 20808730
- [Background] Park YS, Jeon YJ, Kim HS, Han IB, Oh SH, Kim DS, Kim NK. The GC + CC genotype at position -418 in TIMP-2 promoter and the -1575GA/-1306CC genotype in MMP-2 is genetic predisposing factors for prevalence of moyamoya disease. BMC Neurol. 2014 Oct 4;14:180. doi: 10.1186/s12883-014-0180-5. PMID 25280484
- [Background] Perez-Hernandez N, Vargas-Alarcon G, Martinez-Rodriguez N, Martinez-Rios MA, Pena-Duque MA, Pena-Diaz Ade L, Valente-Acosta B, Posadas-Romero C, Medina A, Rodriguez-Perez JM. The matrix metalloproteinase 2-1575 gene polymorphism is associated with the risk of developing myocardial infarction in Mexican patients. J Atheroscler Thromb. 2012;19(8):718-27. doi: 10.5551/jat.11817. Epub 2012 Jun 27. PMID 22785600
- [Background] Sabbatini AR, Barbaro NR, de Faria AP, Ritter AMV, Modolo R, Correa NB, Brunelli V, Pinho C, Fontana V, Moreno H. Matrix metalloproteinase-2 -735C/T polymorphism is associated with resistant hypertension in a specialized outpatient clinic in Brazil. Gene. 2017 Jul 15;620:23-29. doi: 10.1016/j.gene.2017.04.004. Epub 2017 Apr 5. PMID 28390988
- [Background] Strbac D, Goricar K, Dolzan V, Kovac V. Matrix Metalloproteinases Polymorphisms as Prognostic Biomarkers in Malignant Pleural Mesothelioma. Dis Markers. 2017;2017:8069529. doi: 10.1155/2017/8069529. Epub 2017 Sep 12. PMID 29138529
- [Background] Saravani S, Yari D, Saravani R, Azadi Ahmadabadi C. Association of COL4A3 (rs55703767), MMP-9 (rs17576)and TIMP-1 (rs6609533) gene polymorphisms with susceptibility to type 2 diabetes. Biomed Rep. 2017 Mar;6(3):329-334. doi: 10.3892/br.2017.856. Epub 2017 Feb 9. PMID 28451395
- [Background] Chen X, Chen Y, Wiggs JL, Pasquale LR, Sun X, Fan BJ. Association of Matrix Metalloproteinase-9 (MMP9) Variants with Primary Angle Closure and Primary Angle Closure Glaucoma. PLoS One. 2016 Jun 7;11(6):e0157093. doi: 10.1371/journal.pone.0157093. eCollection 2016. PMID 27272641
- [Background] Wu HD, Bai X, Chen DM, Cao HY, Qin L. Association of genetic polymorphisms in matrix metalloproteinase-9 and coronary artery disease in the Chinese Han population: a case-control study. Genet Test Mol Biomarkers. 2013 Sep;17(9):707-12. doi: 10.1089/gtmb.2013.0109. Epub 2013 Jul 2. PMID 23819814
- [Background] Rose BJ, Kooyman DL. A Tale of Two Joints: The Role of Matrix Metalloproteases in Cartilage Biology. Dis Markers. 2016;2016:4895050. doi: 10.1155/2016/4895050. Epub 2016 Jul 13. PMID 27478294
- [Background] Takashiba S, Naruishi K. Gene polymorphisms in periodontal health and disease. Periodontol 2000. 2006;40:94-106. doi: 10.1111/j.1600-0757.2005.00142.x. No abstract available. PMID 16398687
- [Background] Yoon S, Kuivaniemi H, Gatalica Z, Olson JM, Buttice G, Ye S, Norris BA, Malcom GT, Strong JP, Tromp G. MMP13 promoter polymorphism is associated with atherosclerosis in the abdominal aorta of young black males. Matrix Biol. 2002 Oct;21(6):487-98. doi: 10.1016/s0945-053x(02)00053-7. PMID 12392760